CLINICAL TRIAL: NCT05505292
Title: Lifitegrast 5% for the Treatment of Dry Eye In Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Danielle Iacono, Associate Clinical Professor, State University of New York College of Optometry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1449068
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
Keywords: Dry Eye; Soft Contact Lenses
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lifitegrast Ophthalmic Solution Vehicle (Placebo Comparator)
  Interventions: Other: Lifitegrast Ophthalmic Solution Vehicle
- Lifitegrast Ophthalmic Solution 5% (Experimental)
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — Dosed twice a day for 8 weeks
  Other Names: Xiidra
  Arms: Lifitegrast Ophthalmic Solution 5%
Other: Lifitegrast Ophthalmic Solution Vehicle — Dosed twice a day for 8 weeks
  Arms: Lifitegrast Ophthalmic Solution Vehicle

SUMMARY:
This is a prospective, single site, randomized, double masked, comparator-controlled study designed to evaluate the efficacy of lifitegrast ophthalmic solution 5% in treating the symptoms of dry eye in soft contact lens wearers as compared to control. We hypothesize that there will be a significant improvement in dry eye symptoms in contact lens wearers using lifitegrast as compared to those being treated with control (lifitegrast vehicle).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must read, understand and sign the Statement of Informed Consent
2. Subjects must be at least 18 years of age
3. Subjects must be habitual soft contact lens (CL) wearers, with a daily, weekly, bi- weekly or monthly replacement schedule
4. Habitual contact lenses must have a suitable fit as determined by the investigator
5. Subjects must report a history of dry eye symptoms, for which they have used rewetting drops or Artificial Tears (ATs) in the past 30 days
6. Subjects must be willing to discontinue the use of Artificial Tears (ATs) and rewetting drops for the duration of the study
7. Subjects must have a score of 12 or higher on the CLDEQ (Contact Lens Dry Eye Questionnaire-8) at baseline
8. Subjects must have at least 2 of the following signs of dry eye disease:

   1. High tear osmolarity > 308 mOsm/L, (milliosmoles per liter) or a difference greater than 8 mOsm/L between eyes
   2. Any corneal staining
   3. Any bulbar conjunctival staining
   4. Low TBUT (tear break up time) (<10s)
   5. Schirmer <10mm in either eye
9. Subjects must be able to read at least half of the 20/25 (via entrance Snellen visual acuity) or better in each eye in their current contact lens prescription.
10. Subjects currently wearing reusable contact lenses must be willing to use Clear Care solution for cleaning and disinfecting throughout the study.

Exclusion Criteria:

1. Currently pregnant or breastfeeding by self-report
2. Allergy to lifitegrast ophthalmic solution 5% (Xiidra)
3. Habitual extended wear contact lens schedule
4. Any active ocular disease that may affect the ocular surface other than dry eye (significant blepharitis, allergic conjunctivitis, lagophthalmos, chalazia, hordeolum etc.)
5. Any meibomian gland dysfunction, blepharitis, corneal neovascularization or papillary conjunctivitis that is grade 3 or higher using the Efron Grading Scale.
6. Excessive corneal staining, that in the opinion of the investigator, is a contraindication to contact lens use.
7. History of ocular surgery
8. Any active ocular infection
9. Use of any topical ophthalmic medications other than artificial tears or rewetting drops
10. Inability to perform necessary visual function assessments
11. Punctal plug insertion in the last 3 months, or presence of punctal plugs at the time of the exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Iacono, OD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry Clinical Vision Research Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects were enrolled in the study but not randomized due to screen failure
Period: Overall Study
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 subjects who were not randomized due to screenfailure not included
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5% | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.27 (4.57) | 27.20 (5.97) | 26.73 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
CLDEQ8 Total Score [Median (Inter-Quartile Range); unit: units on a scale] — The CLDEQ-8 (Contact Lens Dry Eye Questionnaire) is a symptom questionnaire that assesses discomfort related to dry eye in contact lens wearers. The minimum score (no symptoms) is 0. The maximum score (most symptomatic) is 37. The baseline measure reported is median total score at baseline.
  units on a scale | 21 [19 to 26] | 22 [16 to 24] | 21 [17 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Lifitegrast Ophthalmic Solution 5% in Treating the Symptoms of Dry Eye in Contact Lens Wearers as Measured by Change in Total CLDEQ-8 Score From Baseline to Week 8
Description: Measured by change in total score on the CLDEQ-8 (Contact Lens Dry Eye Questionnaire) in subjects using lifitegrast ophthalmic solution as compared to subjects using lifitegrast ophthalmic solution vehicle from baseline to week 8. The CLDEQ-8 (Contact Lens Dry Eye Questionnaire) is a symptom questionnaire that assesses discomfort related to dry eye in contact lens wearers. The minimum possible CLDEQ-8 score is 0. The maximum possible CLDEQ-8 score is 37. Therefore, the maximum change is +/- 37. A negative change is an improvement in symptoms (a lower score at week 8 than baseline).
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 15
units on a scale | -4 [-8 to -2] | -5 [-8 to -2]
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Total Score on the CLDEQ- 8 From Baseline to 2 Weeks
Description: Measured by change in total score on the CLDEQ-8 (Contact Lens Dry Eye Questionnaire) in subjects using lifitegrast ophthalmic solution as compared to subjects using lifitegrast ophthalmic solution vehicle from baseline to week 2. The CLDEQ-8 (Contact Lens Dry Eye Questionnaire) is a symptom questionnaire that assesses discomfort related to dry eye in contact lens wearers. The minimum possible CLDEQ-8 score is 0. The maximum possible CLDEQ-8 score is 37. Therefore, the maximum change is +/- 37. A negative change is an improvement in symptoms (a lower score at week 2 than baseline).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 15
units on a scale | -3.2 (3.90) | -3.93 (4.96)
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.66, t-test, 2 sided

3. Secondary Outcome: Change in Total Score on the CLDEQ- 8 From Baseline to 4 Weeks
Description: Measured by change in total score on the CLDEQ-8 (Contact Lens Dry Eye Questionnaire) in subjects using lifitegrast ophthalmic solution as compared to subjects using lifitegrast ophthalmic solution vehicle from baseline to week 4. The CLDEQ-8 (Contact Lens Dry Eye Questionnaire) is a symptom questionnaire that assesses discomfort related to dry eye in contact lens wearers. The minimum possible CLDEQ-8 score is 0. The maximum possible CLDEQ-8 score is 37. Therefore, the maximum change is +/- 37. A negative change is an improvement in symptoms (a lower score at week 4 than baseline).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 15
units on a scale | -3.53 (5.18) | -5.6 (3.96)
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.23, t-test, 2 sided

4. Secondary Outcome: Change in Tear Osmolarity OD (Right Eye) From Baseline to Week 8
Description: Change in tear osmolarity (as measured by the TearLab device) from baseline to week 8 in the lifitegrast 5% group compared to subjects using lifitegrast ophthalmic solution vehicle.
  Measured in mOsm/L. A negative change is a lower osmolarity at week 8, which would be an improvement.
Time Frame: 8 weeks
Population: Note that data is missing for 2 subjects in the lifitegrast group due to issues with calibrating the TearLab device on the day of their visits.
Measure: Median (Inter-Quartile Range); unit: mOsm/L (milliosmoles/liter)
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 13
mOsm/L (milliosmoles/liter) | -1 [-14 to 2] | -1 [-11 to 5]
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Tear Osmolarity OS (Left Eye) From Baseline to Week 8
Description: as for outcome 4
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mOsm/L
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 13
mOsm/L | 6 [-11 to 13] | 0 [-12 to 6]
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Forced Choice Questionnaire
Description: Forced choice questionnaire asking if the participant felt that their symptoms improved to the point that they would continue treatment outside of the study
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 15
Participants
  Yes they would continue treatment | 8 | 4
  No they would not continue treatment | 7 | 11
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Test type: Superiority; p = 0.14, Chi-squared

7. Secondary Outcome: Change in Score for Each Question on the CLDEQ-8 From Baseline to Week 8
Description: Measured by change in score for each Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) question in subjects using lifitegrast ophthalmic solution compared to subjects using lifitegrast ophthalmic solution vehicle.
  A negative change for a question from baseline to week 8 is an improvement in symptom frequency or intensity. Questions are for the past 2 weeks.
  Questions 1a, 2a, 3a & 4 ask about frequency of eye discomfort when wearing contacts, eye dryness, changeable, blurry vision in contacts and wanting to close your eyes. Scale: 0=Never, 1=Rarely, 2=Sometimes, 3=Frequently, 4=Constantly Questions 1b, 2b & 3b ask about the intensity of symptoms at the end of contact lens wearing time noted for questions 1a, 2a and 3a. Scale: 0-5, 0=Never have it, 5=Very Intense Question 5 asks how often did your eyes bother you so much that you felt you needed to take out your contact lenses. Scale: 1=Never, 2=Less than once a week, 3=Weekly, 4=Several times a week, 5=Daily, 6=Several times a day
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
Number analyzed (Participants) | 15 | 15
units on a scale
  Question 1A Change | -1 [-2 to 0] | -1 [-1 to 0]
  Question 1B Change | -1 [-2 to 0] | -1 [-2 to -1]
  Question 2A Change | -1 [-1 to 0] | -1 [-1 to 0]
  Question 2B Change | -1 [-1 to 0] | -1 [-1 to 0]
  Question 3A Change | 0 [-1 to 1] | 0 [-1 to 0]
  Question 3B Change | 0 [-1 to 0] | 0 [-2 to 0]
  Question 4 Change | 0 [-1 to 0] | -1 [-1 to 0]
  Question 5 Change | -1 [-1 to 0] | -1 [-2 to -1]
Statistical Analysis 1: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 1a Change from baseline to week 8 in lifitegrast vs vehicle; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 1b change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 2a change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 2b change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 3a change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 3b change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 4 change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Lifitegrast Ophthalmic Solution Vehicle vs Lifitegrast Ophthalmic Solution 5%; Question 5 change from baseline to week 8 in lifitegrast vs vehicle groups; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the 8 weeks of study participation
Arm/Group | Lifitegrast Ophthalmic Solution Vehicle | Lifitegrast Ophthalmic Solution 5%
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast Ophthalmic Solution Vehicle (N=15) | Lifitegrast Ophthalmic Solution 5% (N=15)
Blurry Vision (Eye disorders) | 0 (0) | 2 (2)
Ocular Burning (Eye disorders) | 1 (1) | 3 (3)
Common Cold (Infections and infestations) | 1 (1) | 2 (2)
Conjunctival Hyperemia (Eye disorders) | 1 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Dysguesia (General disorders) | 0 (0) | 7 (7)
Syncope (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Ocular Mucous Discharge (Eye disorders) | 0 (0) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Sore Throat/ Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Stomach Virus (Infections and infestations) | 1 (1) | 0 (0)
Wisdom Tooth Removal (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT05505292/Prot_SAP_000.pdf